CLINICAL TRIAL: NCT02016690
Title: Synagis® Liquid 50mg, 100mg for Intramuscular Injection Special Investigation in Immunocompromised Children With Synagis®
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-296
Record Dates: First submitted 2013-12-11; First posted 2013-12-20 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Prevention of severe RSV infection; Respiratory syncytial virus (RSV) infection; Down Syndrome; Immunocompromised; Effectiveness of palivizumab
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Infections; Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immunocompromised children: Children with immunocompromised conditions or Down syndrome at high-risk of serious RSV disease who received palivizumab during the RSV season

SUMMARY:
This post marketing observational study (PMOS) was conducted in Japan during the 2013-2014 and 2014-2015 Respiratory Syncytial Virus (RSV) seasons to assess the safety and effectiveness of palivizumab for the prevention of serious lower respiratory tract infection caused by RSV in participants 24 months of age and under, who have an immunocompromised medical condition (e.g., combined immunodeficiency disease, antibody deficiency, or other types of immunodeficiency; HIV infection; recovering from organ or bone marrow transplantation; on chemotherapy; on high-dose corticosteroid therapy; on immunosuppressants) or who have Down syndrome.

DETAILED DESCRIPTION:
Palivizumab was prescribed according to the local label and independently of the decision to enroll participants in the study. Palivizumab was administered monthly throughout the Respiratory Syncytial Virus (RSV) infection seasons via intramuscular injection at a dose of 15 mg/kg of body weight. Survey forms were collected after the observation period. The number of adverse events and the frequency of hospitalizations due to RSV infections in surveyed participants were assessed to evaluate the safety and effectiveness of palivizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of a parent or legal guardian who was capable and willing to give written informed consent for his/her newborn, infant or young child to participate in the study
2. Participants receiving palivizumab for prevention of serious lower respiratory tract disease caused by RSV infection
3. Newborns, infants, or young children 24 months of age and under who have an immunocompromised medical condition:

   * combined immunodeficiency, (severe combined immunodeficiency, X-linked hyper-immunoglobulin M (IgM) syndrome, etc.), antibody deficiency (X-linked agammaglobulinemia,common variable immunodeficiency, non-X-linked hyper-IgM syndrome,etc.) or other immunodeficiency (Wiskott-Aldrich syndrome, etc.)
   * acquired T cell dysfunction ( such as human immunodeficiency virus (HIV) infection etc.)
   * history of past organ transplantation
   * history of past bone marrow transplantation
   * receiving immunosuppressive chemotherapy
   * receiving systemic high-dose corticosteroid therapy (prednisone equivalents ≥ 0.5 mg/kg/every other day, other than inhaler or topical use), or
   * receiving other immunosuppressive therapy (azathioprine, methotrexate, mizoribine, mycophenolate mofetil, cyclophosphamide, cyclosporine, tacrolimus, cytokine inhibitors, etc.)
   * receiving biologics (including cytokine inhibitors)
   * Others (nephrotic syndrome, chronic peritoneal dialysis, hemodialysis)
4. Newborns, infants, or young children age of 24 months and under who have Down syndrome without a current hemodynamically significant Congenital Heart Disease. The participant must have had an experience with persistent respiratory symptoms or regular outpatient treatment due to respiratory tract infection prior to current RSV season.

Exclusion criteria:

1. Participants included in the Contraindications section of the package insert
2. Participants with known hypersensitivity to the ingredients of palivizumab
3. Participants with a known positive RSV infection before hospitalization

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Single-arm, Multi-center, Prospective Cohort
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Mikami, MD, PhD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled via consecutive enrollment method who had a completed CRF. Participants were excluded if there was enrollment at a non-contracting institution or beyond the contracted number; duplicate enrollment; no palivizumab administration; or if palivizumab administration began outside of the investigation period.
Period: Overall Study
Arm/Group | Immunocompromised Children
Started | 312
Treated | 312
Safety Analysis Set (SAS) | 304
Completed | 288 ((Effectiveness analysis set))
Not Completed | 24
Not completed — Excluded from SAS: Enrollment violation | 2
Not completed — Excluded from SAS: Duplication | 2
Not completed — Excluded from SAS: Early treatment | 2
Not completed — Excluded from SAS: Ineligible for study | 2
Not completed — Did not meet inclusion criteria | 13
Not completed — Hospitalized for RSV at study start | 3

BASELINE CHARACTERISTICS:
Population: Participants enrolled via consecutive enrollment method who had a completed CRF. Participants were excluded if there was enrollment at a non-contracting institution or beyond the contracted number; duplicate enrollment; no palivizumab administration; or if palivizumab administration began outside of the investigation period.
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 304
Age, Continuous [Mean (Standard Deviation); unit: months] | 11.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 297
  Black | 0
  White | 0
  Asian | 3
  Others | 4
Age at the start of treatment [Count of Participants; unit: Participants]
  ≤ 1 month | 31
  > 1 and ≤ 3 months | 24
  > 3 and ≤ 6 months | 31
  > 6 and ≤ 12 months | 81
  > 12 and ≤ 24 months | 137
  > 24 months | 0
Body weight at the start of treatment [Count of Participants; unit: Participants]
  < 1000 grams | 0
  ≥ 1000 and < 1500 grams | 0
  ≥ 1500 and < 2500 grams | 1
  ≥ 2500 and < 5000 grams | 52
  ≥ 5000 and < 10000 grams | 202
  ≥ 10000 and < 15000 grams | 45
  ≥ 15000 grams | 1
  Not specified | 3
Gestational age [Count of Participants; unit: Participants]
  < 22 weeks | 0
  ≥ 22 and < 37 weeks | 56
  ≥ 37 and < 42 weeks | 237
  ≥ 42 weeks | 1
  Not specified | 10
Body weight at birth [Count of Participants; unit: Participants]
  < 1000 grams | 0
  ≥ 1000 and ≤ 1500 grams | 4
  ≥ 1500 and ≤ 2500 grams | 80
  ≥ 2500 and ≤ 4000 grams | 207
  ≥ 4000 grams | 2
  Not specified | 11
Number of smokers in the household [Count of Participants; unit: Participants]
  0 smokers | 184
  ≥ 1 smokers | 40
  Not specified | 80
Familial predisposition to hypersensitivity [Count of Participants; unit: Participants]
  No | 180
  Yes | 34
  Unknown | 84
  Not specified | 6
Participant's predisposition to hypersensitivity [Count of Participants; unit: Participants]
  No | 245
  Yes- asthma | 11
  Yes- allergic bronchitis | 1
  Yes- allergic rhinitis | 4
  Yes- allergic dermatitis | 4
  Yes- food allergy | 11
  Yes- drug allergy | 3
  Yes- others | 1
  Unknown | 28
Comorbidity [Count of Participants; unit: Participants]
  No | 120
  Yes- renal disease | 18
  Yes- hepatic disease | 21
  Yes- respiratory disease | 50
  Yes- cardiovascular disease | 45
  Yes- others | 142
  Unknown | 1
Lower Respiratory Tract Infection score at the start of treatment [Count of Participants; unit: Participants] — The Lower Respiratory Tract Infection (LRI) Score ranged from 0 (well or baseline); 1(Upper Respiratory tract Infection [URI]), mild; 2 (LRI); 3 (LRI, moderate); 4 (LRI, severe) to 5 (Respiratory Failure). Components of the score included respiratory rate per minute, oxygen saturation, and physical findings. LRI scores were documented on the case report form (CRF).
  Participants
    0 | 289
    1 | 5
    2 | 4
    3 | 4
    4 | 1
    5 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with their treatment. Adverse events were documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 304
Participants | 99

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event was defined as any untoward medical occurrence in a participant that the investigator believed to be causally related to the study treatment and met at least one of the following criteria: death, life-threatening, hospitalization or prolongation of hospitalization, persistent or significant disability/incapacity, or important medical event requiring medical or surgical intervention to prevent serious outcome. Serious adverse events were documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 304
Participants | 53

3. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with their treatment. If a causal relationship with palivizumab was: "Related", "Causality cannot be ruled out", or "Not assessable" as determined by the investigator, it was classified as an adverse drug reaction (ADR). An AE was considered a serious adverse event (SAE) and a serious adverse drug reaction (SADR) if the severity of the AE or ADR was any one of the following, as determined by the investigator: "Death", "Life-threatening condition", "Hospitalization or prolonged hospitalization", "Persistent or significant disability", or "Other medically important condition". Information about AEs and ADRs was documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 304
Participants | 25

4. Secondary Outcome: Change in Lower Respiratory Tract Infection (LRI) Score During the Study
Description: The Lower Respiratory Tract Infection (LRI) Score ranged from 0 (well or baseline); 1 (Upper Respiratory tract Infection [URI]), mild); 2 (LRI); 3 (LRI, moderate); 4 (LRI, severe) to 5 (Respiratory Failure). Components of the score included respiratory rate per minute, oxygen saturation, and physical findings of LRI. LRI scores were documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab up to the last administration of palivizumab, up to 36 weeks
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 288
units on a scale
  1 dose | 0.1 (0.6)
  2 doses: number analyzed (Participants) | 254
  2 doses | 0.1 (0.6)
  3 doses: number analyzed (Participants) | 231
  3 doses | 0.1 (0.6)
  4 doses: number analyzed (Participants) | 213
  4 doses | 0.1 (0.6)
  5 doses: number analyzed (Participants) | 192
  5 doses | 0.1 (0.4)
  6 doses: number analyzed (Participants) | 159
  6 doses | 0.1 (0.3)
  7 doses: number analyzed (Participants) | 126
  7 doses | 0.0 (0.2)
  8 doses: number analyzed (Participants) | 54
  8 doses | 0.1 (0.3)
  9 doses: number analyzed (Participants) | 3
  9 doses | 0.0 (0.0)

5. Secondary Outcome: Number of Participants Hospitalized Due to Respiratory Syncytial Virus (RSV) Infection
Description: Hospitalization due to RSV infection or the presence/absence of positive RSV antigen test results during hospitalization was documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 5
Participants | 2

6. Secondary Outcome: Mean Hospitalization Length Due to Respiratory Syncytial Virus (RSV) Infection
Description: The date of hospitalization due to RSV infection and the date of hospital discharge were documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 2
days | 9.5 (2.1)

7. Secondary Outcome: Number of Hospitalized Participants Requiring Respiratory Support
Description: The presence/absence of respiratory support, (oxygen therapy, mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure, and other mechanical respiratory support or Intensive Care Unit admission) the start and end dates of respiratory support, and the dates of hospitalization and discharge were documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 2
Participants | 1

8. Secondary Outcome: Mean Duration of Respiratory Support
Description: The presence/absence of respiratory support (oxygen therapy, mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure, and other mechanical respiratory support or Intensive Care Unit admission) and the start and end dates of respiratory support were documented on the case report form (CRF).
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab, up to 44 weeks
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Immunocompromised Children
Number analyzed (Participants) | 3
days | 40.0 (62.4)

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of study drug administration until 30 days after the last dose of study drug, up to 44 weeks.
Arm/Group | Immunocompromised Children
Serious Adverse Events (participants affected / at risk) | 53/304
Other Adverse Events (participants affected / at risk) | 67/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunocompromised Children (N=304)
Bacteraemia (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 3
Cytomegalovirus infection (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 2
Respiratory syncytial virus infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 3
Chronic graft versus host disease (Immune system disorders) | 2
Adrenal disorder (Endocrine disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Febrile convulsion (Nervous system disorders) | 2
Neurological symptom (Nervous system disorders) | 1
Eyelid oedema (Eye disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Hypertension (Vascular disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Anal atresia (Congenital, familial and genetic disorders) | 1
X-linked lymphoproliferative syndrome (Congenital, familial and genetic disorders) | 1
Omenn syndrome (Congenital, familial and genetic disorders) | 1
Condition aggravated (General disorders) | 1
Pyrexia (General disorders) | 2
Neutrophil count decreased (Investigations) | 1
Norovirus test positive (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunocompromised Children (N=304)
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 3
Croup infectious (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Exanthema subitum (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 3
Enteritis infectious (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 2
Enterocolitis viral (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Viral rhinitis (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Metapneumovirus infection (Infections and infestations) | 1
Tinea manuum (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 2
Engraftment syndrome (Immune system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1
Epilepsy (Nervous system disorders) | 1
Uveitis (Eye disorders) | 1
Hypertension (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 22
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Enterocolitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Alanine aminotransferase increased (Investigations) | 1
Blood culture positive (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 1
Antithrombin III decreased (Investigations) | 1
Aspergillus test positive (Investigations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Frostbite (Injury, poisoning and procedural complications) | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study population was a very specific, defined group, observed in the context of daily practice.The results of this study of the safety and effectiveness of palivizumab may not be applicable to the general population of healthy infants in Japan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.